CLINICAL TRIAL: NCT04825535
Title: A Non-Inferiority Randomized Controlled Trial Comparing Online and On-Site Cognitive Behaviour Therapy in Major Depressive Disorder
Brief Title: Non-Inferiority RCT Comparing Online and On-Site CBT in MDDi
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study suspended due to issues flagged during an internal Quality Assurance audit.
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-2020
Record Dates: First submitted 2021-03-21; First posted 2021-04-01 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Major Depressive Disorder
Keywords: internet-based intervention; major depressive disorder; health coaching
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Online CBT intervention
Who Masked: Outcomes Assessor
Masking Description: One assessor will be blinded to the (2) comparison groups of all participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard psychiatry and cognitive behavioural online intervention (Experimental): The online group CBT-M program combines software-based workbooks with phone-based Navigator-Coaching that coordinates software interactions (e.g., secure text messaging, Fitbit tracked walking, food monitoring via photography). Navigation coaching is supplied by students who were pursuing graduate degrees (MSc, MA, PhD) in kinesiology and health science, education, and psychology.
  Interventions: Behavioral: Standard psychiatry and cognitive behavioral online intervention
- Standard psychiatry and cognitive behavioural in-person intervention (Active Comparator): The on-site, usual-care CBT group follows the structure of the Mind Over Mood workbook in reviewing CBT concepts and procedures. A series of work sheets assist participants in differentiating moods, and in differentiating moods from thoughts and situational influences, leading to modifications of thinking, behaviour, emotion and mood. Group leaders are standard leaders in the CAMH group-CBT program who have Masters-level degrees in psychology, social work and occupational therapists.
  Interventions: Behavioral: Standard psychiatry and cognitive behavioural in-person intervention

INTERVENTIONS:
Behavioral: Standard psychiatry and cognitive behavioral online intervention — The cognitive behavioral online intervention has been assessed in a prior trial. Ritvo, P, Knyahnytska, Y, Pirboglou, M, Wang, W, Tomlinson, G, Zhao, H, Linklater, R, Kirk, M., Katz, J., Harber, L., Daskalakis, ZJ An online mindfulness-based cognitive behavioural therapy intervention for youth diagnosed with major depressive disorders: J Med Internet Res 2021, Mar 17; 23 (3), e24380
  Arms: Standard psychiatry and cognitive behavioural online intervention
Behavioral: Standard psychiatry and cognitive behavioural in-person intervention — The effectiveness of standard care office-based group CBT-MM at CAMH is indicated in a past study (n = 119) where depression symptoms reduced (after 16 weeks treatment) by 27% [3,18 ]. The office-based groups follow a carefully conceived structure that centers on the workbook Mind Over Mood (MOM) (Guilford Press) [41]. Key CBT concepts and procedures are conveyed via work sheets that structure personal and group exploration.
  Arms: Standard psychiatry and cognitive behavioural in-person intervention

SUMMARY:
In recent years, Cognitive Behavioral Therapy has been integrated with mindfulness meditation (CBT-M) following evidence for increased efficacy when modalities are combined. We will assess whether online group CBT-M plus standard psychiatric care is non-inferior in efficacy and more cost-effective than office-based, on-site group CBT-M (plus standard psychiatric care) per outcomes at post-intervention and at 6-month follow up in adults with major depressive disorder (MDD). This non-inferiority randomized controlled trial will employ both assessor-blinded and self-report outcome measures and will include a full economic evaluation.

DETAILED DESCRIPTION:
Depression is a commonly diagnosed mental health disorder that represents the most prevalent cause of disability worldwide. Cognitive Behavioural Therapy (CBT) is the best-evidenced treatment for depression, but despite demonstrated efficacy, many individuals cannot access adequate psychotherapeutic treatment due to the limitations of face-to-face delivery. In recent years, CBT has been integrated with mindfulness meditation (CBT-M) following strong evidence for increased efficacy when the two modalities are combined. Previous RCTs have demonstrated that online CBT-M is effective in depressive symptom reduction, but direct comparisons to in-office CBT delivery assessing cost and treatment outcomes are required to facilitate innovation and clinical policy change.

Objectives: To assess whether online group CBT-M plus standard psychiatric care is non-inferior in efficacy and more cost-effective than office-based, on-site group CBT-M (plus standard psychiatric care) per outcomes at post-intervention and at 6-month follow up in adults diagnosed with major depressive disorder (MDD). The study will assess whether digitally recorded adherence data (i.e. online workbooks completed, Fitbit tracked step count, online text-messages exchanged, phone sessions completed) predict outcome benefits in the online-group participants as measured by changes in depressive symptoms.

Methods: This single-centre, 2-arm non-inferiority randomized controlled trial will employ both assessor-blinded and self-report outcome measures and will include a full economic evaluation.

The research site is the Centre for Addiction and Mental Health (CAMH), a large research-based psychiatry institution located in Toronto, Canada. Participants will be identified from wait-lists for CAMH services and through contacts with other Toronto outpatient clinics.

Interventions: All participants will receive standard psychiatric care (1 pharmacotherapy focused visit/month with a psychiatrist of 15-30 minute duration). Experimental participants additionally receive online CBT-M while control participants receive standard care in-office group CBT-M. The online group CBT-M program (in collaboration with NexJ Health, Inc.) combines exposure to smartphone and computer accessed workbooks with phone-based mental health counselling (16 hours in 16 weeks) that coordinates with ongoing software interactions (e.g. secure text messaging, Fitbit tracked walking). Each participant is loaned a Fitbit-HR Charge 3 to assess physical activity as measured by daily step count.

ELIGIBILITY:
Inclusion Criteria:

* Beck Depression Inventory-II of at least mild severity (BDI-II score ≥ 14) with no upper severity limit;
* Psychiatrist diagnosis of Major Depression Disorder;
* Mini-International Neuropsychiatric Interview (MINI)-confirmed diagnosis of Major Depression Disorder;
* fluent in English.

Exclusion Criteria:

* individuals currently receiving weekly structured psychotherapy;
* individuals who meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) criteria for severe alcohol/substance use disorder (in the past 3 months), borderline personality disorder, schizophrenia or any other primary psychotic disorder, bipolar disorder or obsessive-compulsive disorder;
* individuals who manifest clinically significant suicidal ideation defined as imminent intent or attempted suicide (in the past 6 months);
* individuals who are judged to have treatment resistant depression (TRD), as defined by failure in at least two trials of antidepressant medications and/or a course of psychotherapy during the current depressive episode

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 156 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change in Beck Depression Inventory - 2 (0 to 63 - higher score indicates worse outcome) | Baseline and 4 months
  Frequently used and validated self report measure

SECONDARY OUTCOMES:
Change in Beck Anxiety Inventory (0 to 63 - higher score indicates worse outcome) | Baseline and 4 months
  Frequently used and validated self report measure
Change in Quick Inventory of Depressive Symptoms (0 to 48 - higher score indicates worse outcome) | Baseline and 4 months
  Frequently used and validated self report measure
Change in Hamilton Depression Rating Scale - 24-item version (0 to 72) Hamilton Depression Rating Scale - 24 item (0 - 96 - higher score indicates worse outcome) | Baseline and 4 months
  Frequently used and validated interview-based evaluation instrument
Change in 5-Facet Mindfulness Questionnaire - 39-item version (39 to 195 - higher score indicates better outcome) Five-Facet Mindfulness Questionnaire | Baseline and 4 months
  Frequently used and validated self report measure
Change in Brief Pain Inventory - 11 item (0 - 176 - high score indicates worse outcome) | Baseline and 4 months
  Frequently used and validated self report measure
Change in EuroQol-5 Dimension (EQ-5D) Quality of Life Instrument - 5 items - 0 - 25 - high score - worse outcome) | Baseline and 4 months
  Frequently used and validated self report measure

CONTACTS AND LOCATIONS:
Overall Officials: David Gratzer, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No. We may consider investigators who wish to use data in further analyses but we cannot guarantee access.

REFERENCES:
- [Derived] Ritvo P, Gratzer D, Knyahnytska Y, Ortiz A, Walters C, Katz J, Laposa J, Baldissera C, Wayne N, Pfefer-Litman D, Tomlinson G, Daskalakis Z. Comparing Online and On-Site Cognitive Behavior Therapy in Major Depressive Disorder: Protocol for a Noninferiority Randomized Controlled Trial. JMIR Res Protoc. 2022 Apr 8;11(4):e29726. doi: 10.2196/29726. PMID 35393942